CLINICAL TRIAL: NCT04416568
Title: Phase 2 Proof of Concept Study of Nivolumab and Ipilimumab in Children and Young Adults With Relapsed or Refractory INI1-negative Cancers
Brief Title: Study of Nivolumab and Ipilimumab in Children and Young Adults With INI1-Negative Cancers
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Gateway for Cancer Research (Other)
Responsible Party: Principal Investigator, Suzanne Forrest, MD, Sponsor Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-041
Record Dates: First submitted 2020-06-02; First posted 2020-06-04 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Malignant Rhabdoid Tumor; Rhabdoid Tumor of the Kidney; Epithelioid Sarcoma; Chordoma (Poorly Differentiated or De-differentiated); Atypical Teratoid/Rhabdoid Tumor; Other INI1 Negative Tumors (With PI Approval); Other SMARCA4-deficient Malignant Tumors (With PI Approval)
Keywords: Malignant Rhabdoid Tumor; Rhabdoid Tumor of the Kidney; Epithelioid Sarcoma; Chordoma (poorly differentiated or de-differentiated); Atypical Teratoid/Rhabdoid Tumor; INI1 negative tumors; SMARCA4-deficient malignant tumors
MeSH Terms: conditions — Rhabdoid Tumor; Sarcoma; Chordoma | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Solid Tumor (Stratum 1) (Experimental): * Patients will receive combination therapy with nivolumab at a predetermined dose and ipilimumab at a predetermined dose day 1 of a 21-day cycle for 4 cycles
  * Starting with cycle 5, patients will receive nivolumab monotherapy at a predetermined dose on day 1 and day 15 of a 28-day cycle
  * Patients with INI1-negative relapsed or refractory extracranial solid tumors
  Interventions: Drug: Nivolumab; Drug: Ipilimumab
- CNS (Stratum 2) (Experimental): * Patients will receive combination therapy with nivolumab at a predetermined dose and ipilimumab at a predetermined dose day 1 of a 21-day cycle for 4 cycles
  * Starting with cycle 5, patients will receive nivolumab monotherapy at a predetermined dose on day 1 and day 15 of a 28-day cycle
  * Patients with INI1-negative relapsed or refractory CNS tumors
  Interventions: Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: Nivolumab — Combination Therapy: Nivolumab at predetermined dosage day 1 of a 21-day cycle for 4 cycles.
  Monotherapy: Starting with cycle 5 nivolumab at predetermined dosage on day 1 and day 15 of a 28-day cycle
  Other Names: OPDIVO
Drug: Ipilimumab — Combination Therapy: Ipilimumab at predetermined dosage day 1 of a 21-day cycle for 4 cycles
  Other Names: YERYOY

SUMMARY:
This clinical trial is studying two immunotherapy drugs (nivolumab and ipilimumab) given together as a possible treatment for INI1-negative tumors.

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial, which tests the safety and effectiveness of an investigational drug or drug combination to learn whether the drug or drug combination works in treating a specific disease. "Investigational" means that the drug combination is being studied.

The names of the study drugs involved in this study are:

* Nivolumab (OPDIVO)
* Ipilimumab (YERYOY)

This trial is studying whether nivolumab and ipilimumab work to treat INI1-negative cancers.

The U.S. Food and Drug Administration (FDA) has not approved combination nivolumab and ipilimumab for the specific diseases in this study but it has been approved for other diseases. Nivolumab and ipilimumab have been tested in children to find out a safe dose of this combination.

ELIGIBILITY:
Inclusion Criteria:

* All participants must have one of the following histologically confirmed tumors at original diagnosis or relapse:

  * Stratum 1

    * Malignant rhabdoid tumor (MRT)
    * Rhabdoid tumor of the kidney (RTK)
    * Epithelioid sarcoma
    * Chordoma (poorly differentiated or de-differentiated)
    * Other INI1-negative or SMARCA4-deficient malignant tumors (with PI approval)
  * Stratum 2

    * Atypical teratoid rhabdoid tumor (ATRT)
    * Other INI1-negative or SMARCA4-deficient primary CNS malignant tumors (with PI approval)
* All participants must have tumor assessment at original diagnosis or relapse showing the following:

  * Loss of INI1 confirmed by immunohistochemistry (IHC), OR
  * Molecular confirmation of tumor bi-allelic SMARCB1 (INI1) loss or mutation when INI1 IHC is equivocal or unavailable
  * Loss of SMARCA4 confirmed by IHC or molecular confirmation of tumor bi-allelic SMARCA4 loss or mutation when SMARCA4 is equivocal or unavailable
* Relapsed or refractory disease and no standard treatment options as determined by locally or regionally available standards of care and treating physician's discretion
* Measurable disease as defined by RECIST v1.1 (Stratum 1) or RANO criteria (Stratum 2)
* Karnofsky performance status ≥ 50% for participants ≥16 years of age and Lansky performance status ≥ 50% for participants <16 years of age
* Participants must have fully recovered from the acute toxic effects of all prior anti-cancer therapy. Participants must meet the following minimum washout periods prior to first day of study treatment:

  * Myelosuppressive chemotherapy: At least 14 days after the last dose of myelosuppressive chemotherapy
  * Radiotherapy

    * At least 14 days after local palliative XRT (small port)
    * At least 90 days must have elapsed after prior TBI, craniospinal XRT or if >50% radiation of pelvis
    * At least 42 days must have elapsed if other substantial BM radiation
    * At least 42 days must have passed since last radionuclide therapy (e.g. samarium or radium)
  * Small molecule biologic therapy: At least 7 days following the last dose of a nonmonoclonal biologic agent
  * Monoclonal antibody: At least 21 days after the last dose
  * Myeloid growth factors: At least 14 days following the last dose of long-acting growth factor (e.g. Neulasta) or 7 days following short-acting growth factor
  * Stem Cell or Autologous T Cell Infusion: At least 42 days must have elapsed after stem cell or autologous T cell infusion
* Participants must have adequate organ function as defined below

  * Bone Marrow Function

    * Absolute neutrophil count ≥500/uL
    * Platelets ≥50,000/uL and transfusion independent
  * Hepatic Function

    * Total bilirubin ≤ 1.5 x upper limit of normal for age
    * ALT (SGPT) ≤ 3 x upper limit of normal
  * Renal function

    * A serum creatinine within protocol limits based on age/sex. OR
    * Creatinine clearance ≥ 70 mL/min/1.73 m2 for participants with creatinine levels above institutional normal
  * Adequate Pulmonary Function Defined as: no evidence of dyspnea at rest, no exercise intolerance due to pulmonary insufficient and a pulse oximetry > 92% while breathing room air
  * Adequate pancreatic function defined as serum lipase ≤ ULN at baseline
  * Negative B-HCG pregnancy test in females of childbearing potential (must be drawn within 24 hours prior to initial administration of nivolumab)
  * Women of childbearing potential (WOCBP) receiving nivolumab agree to adhere to contraception for a period of 5 months after the last dose of nivolumab. Men receiving nivolumab and who are sexually active with WOCBP will agree to adhere to contraception for a period of 7 months after the last dose of nivolumab.
  * Ability to understand and/or the willingness of the patient (or parent or legally authorized representative, if minor) to provide informed consent using an institutionally approved informed consent procedure.

Exclusion Criteria:

* Participants who are receiving any other investigational agents.
* Participants must not be receiving concomitant systemic steroid medications The use of physiologic doses of corticosteroids (up to 5 mg/m2/day prednisone equivalent) may be approved after consultation with the PI (treatment with topical, inhaled or ophthalmic corticosteroid is acceptable)
* Participants with a known history of HIV, hepatitis B, and/or hepatitis C
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or any other concurrent disease which in the judgment of the Investigator would make the subject inappropriate for enrollment on this study
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis
* Has active autoimmune disease that has required systemic treatment in the past 12 months, or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo or resolved childhood asthma/atopy are exceptions. Intermittent use of bronchodilators or local steroid injections are not excluded. Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. Autoimmune diagnoses not listed must be approved by the Principal Investigator.
* Patients who have received prior solid organ transplantation are not eligible.
* Pregnancy or Breast-Feeding. Pregnant or breast-feeding women will not be entered on this study due to risks of fetal and teratogenic adverse events as there is yet no available information regarding human fetal or teratogenic toxicities. Pregnancy tests must be obtained in girls who are post-menarchal.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2 or anti-CTLA4 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g. OX-40, CD137)
* Participants who have received live / attenuated vaccine within 30 days of first dose of study treatment.

Ages: 6 Months to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Estimated)
Dates: Start 2020-08-14 (Actual); Primary Completion 2025-07-17 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Objective Overall Response Rate (Stratum 1) | 12 months
  Based on Response Evaluation in Solid Tumors (RECIST) version 1.1
Objective Overall Response Rate (Stratum 2) | 12 months
  Based on Response Assessment in Neuro-Oncology (RANO) Criteria

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 3 years
  Time from study enrollment until the first occurrence of disease progression, relapse or death due to disease
Overall survival (OS) | 3 years
  Time from study enrollment until death from any cause
Disease control rate at 12 months | 12 Months
  The proportion of patients who are progression-free at 12 months
Occurrence of toxicities (Grade 3-5 per CTCAE) | 13 months
  Assessed by National Cancer Institute Common Terminology Criteria for Adverse Events, version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Forrest, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (8):
- United States (8):
  - UCSF Benioff Children's Hospital, San Francisco, California
  - Children's Healthcare of Atlanta-Egleston, Atlanta, Georgia
  - Children's Healthcare of Atlanta-Scottish Rite, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu